CLINICAL TRIAL: NCT06878092
Title: Feasibility and Acceptability of Problem Management Plus With Emotional Processing (PM+EP) for Forcibly Displaced Youth Living in Sweden
Brief Title: Problem Management Plus With Emotional Processing (PM+EP) for Forcibly Displaced Youth
Acronym: PM+EP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Rädda Barnen (Unknown)
Responsible Party: Principal Investigator, Aemal Akhtar, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-05883-02
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Psychological Distress; Traumatic Stress
Keywords: psychological distress; scalable psychological interventions; forcibly displaced; common mental disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Problem Management Plus with Emotional Processing (PM+EP) (Experimental)
  Interventions: Behavioral: Problem Management Plus with Emotional Processing Module (PM+EP)
- Problem Management Plus (Active Comparator)
  Interventions: Behavioral: Problem Management Plus (PM+)
- Treatment as Usual (Other)
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — Problem Management Plus is a brief, potentially scalable psychological intervention developed by the World Health Organization and is delivered by non-specialised helpers. In brief, the intervention is based on cognitive behavioural therapy (CBT) techniques and typically consists of five weekly, ninety-minute sessions. Participants are taught the following techniques during the sessions: stress management, problem-solving, behavioural activation, and accessing social support. The effectiveness of both the individual and group formats of the PM+ intervention have been shown in a number of large definitive RCTs. For the purposes of this study, an adapted version of PM+ will be used to match the exposure between the two active intervention arms. There will be six, weekly seventy-five-minute sessions
  Arms: Problem Management Plus
Behavioral: Problem Management Plus with Emotional Processing Module (PM+EP) — To more directly address symptoms of traumatic stress, an adapted version of PM+ containing Emotional Processing module will be trialed in this study. The PM+ strategies discussed above are identical across both interventions apart from the additional module. The Emotional Processing module aims to provide a safe environment for participants to engage in the emotional processing of both positive and negative memories. During the additional session, participants will be asked to imagine significant memories as pieces of a jigsaw puzzle; participants will be asked to illicit three memories, two positive/pleasurable and one negative/frightening. Participants will be assisted in processing these memories through discussing the puzzle pieces, the thoughts and emotions that come with the memory, and future perspectives. Participants will be asked to rate the intensity of emotions before and after they talk about their memories each time they are brought up.
  Arms: Problem Management Plus with Emotional Processing (PM+EP)
Other: Care as usual — The comparison group will receive care as usual (CAU) only. CAU for forcibly displaced youth (under 18) in Sweden corresponds to primary health care, education, social protection services, and specialized psychological treatment programs. However, adults are only able to access care that cannot be deferred. Once the individual has received their residence permit, they are able to access all healthcare. Upon first arriving in Sweden, refugees are referred to a municipality by the Swedish Board of Migration (Migrationsverket) until they have their residence permit. The municipality is responsible for education and social services while the regions are responsible for health care. In the regions, primary care is responsible for the first line of treatment but can also refer to the child and adolescent mental health services (CAMHS) if needed. Unaccompanied children might either be placed in families or in residential facilities and benefit from the same systems as accompanied children.
  Arms: Treatment as Usual

SUMMARY:
The goal of this feasibility randomized controlled trial is to learn about the feasibility and acceptability of scalable psychological interventions in Sweden. It will also allow for a preliminary exploration of a novel modular addition targeting traumatic stress to Problem Management Plus (PM+), an evidence-based transdiagnostic psychological intervention for psychological distress.

The main question it aims to answer is whether PM+ and PM+ Emotion Processing (PM+EP) feasible and acceptable among forcibly displaced youth in Sweden?

Participants will be randomized to receive PM+, PM+EP, or treatment as usual. The two intervention arms consist of a weekly session for six weeks.

Assessments will collect data on a variety of psychological symptoms, wellbeing, and service use throughout the duration of the study. Assessments will take place at baseline, 1-week post-intervention, and 3-weeks post-intervention.

DETAILED DESCRIPTION:
Study Procedure

Potential participants will be approached through Save the Children and other non-government organizations (NGOs), varied community sources, including service providers, and social media. Given the locations of Save the Children activities, in-person recruitment efforts through will primarily focus on Stockholm, Malmo, and Gothenburg regions. All participants will provide oral and written informed consent, either in Swedish or in their native language, depending on preference, prior to taking part in the screening process. For participants aged 16 - 17, the individuals will be asked to provide contact details to their parents before assessment to make sure that we can contact the parents in case of that the child describes severe symptoms such as suicidal ideation at the assessment. The participants will also get written information about the study to provide to their parents. For potential participants with literacy difficulties, a witnessed thumb print will be collected in lieu of written consent, according to WHO guidelines. Prior to participation, it will be ensured that consenting participants are fully aware of what it means to participate in the trial and that they have the autonomy to withdraw their consent at any time without having to give an explanation. It will also be made abundantly clear that for those who refuse to participate, it will not have an impact on any other types of support that they may be receiving or have access to in the community through community and non-governmental organization initiatives. Consenting participants will be invited to complete self-report screening assessments which includes the capture of basic socio-demographic data and the following measures: K10, WHODAS 2.0, and WHO PM+ suicide screening tool. Following the screening procedures, an assessor will determine whether the participants met the inclusion or exclusion criteria. For participants who did not screen positive for psychological distress, assessors will provide them with feedback indicating that they are dealing with their stress in a healthy manner; if participants express further concern, they will be informed of resources on available services and psychosocial support options in their communities. Those who are excluded due to meeting one of the exclusion criteria, indicative of more severe problems, will be referred to child- and adolescent or adult psychiatric services, depending on their age.

Eligible participants will be invited to participate in the trial and to complete a baseline assessment either live or by teleconferencing (Table 1). Participants will complete measures examining the following constructs: anxiety and depression (Hopkins Symptom Checklist-25; HSCL-25), PTSD (PTSD Checklist for DSM-5; PCL-5), self-identified problems (Psychological Outcomes Profile; PSYCHLOPS), well-being (WHO-5 Well-being Index; WHO-5), social support, agency (State Hope Scale for Adolescents; SHS-A), and health care services recently received (Client Service Receipt Inventory; CSRI). In addition, participants will complete checklists indicating pre- and post-migration stressors. All screening and baseline assessments will be completed during Save the Children work hours (08:00 - 16:00) to ensure that appropriate referrals are able to be made according to their standard operating procedures if imminent risk of suicide is expressed during the assessments. Following the completion of the baseline assessment, participants will be randomized as described in detail below.

Following randomization, if participants are to receive the PM+ or PM+EP intervention, they will be contacted by either a PM+ or PM+EP facilitator who will schedule the upcoming six sessions. If participants are to receive CAU, they will receive a phone call from a Save the Children employee and be referred to Save the Children's programs/other programmes locally providing psychosocial care. Following both the completion of the baseline assessments and randomization, participants will be contacted to organize the first session within seven days. The first session will take place no longer than two weeks following the baseline assessments. Participants will be given the choice as to whether they prefer the PM+/PM+EP intervention to be provided in-person or through teleconferencing. If during the study there are any COVID-19/pandemic related restrictions or other reasons stated by the participants that require remote administration of the intervention, teleconferencing will be used. The post-intervention assessment will take place within two weeks after completion of the sixth and final session (participants can take up to 11 weeks to complete six sessions). The post-assessments will include the WHODAS 2.0, HSCL-25, PCL-5, PSYCHLOPS, CSRI, WHO-5, social support, and SHS-A assessments. The follow-up assessment will be conducted three months after the sixth PM+ session (i.e. 18 weeks after baseline). The assessment will be identical to the post-intervention assessment but will additionally include the checklists that were collected during the baseline assessments.

Randomisation

Randomisation will be conducted by an independent researcher not involved in the study following the participants completion of the baseline assessment. The randomization sequence will be generated by electronic software with a 1:1:1 allocation ratio between PM+, PM+EP, and CAU; randomization will be stratified by participant language and region of recruitment. Following randomization, the participant will be connected with either a PM+ or PM+EP helper, or CAU facilitators who will then independently plan the upcoming intervention schedule. As this is a single-blind RCT, the assessors who will collect pre-, post-, and follow-up data will not be aware of which form of PM+ participants received during their treatment and where possible a different assessor will conduct each of the three assessments for a given participant. For follow-up assessments, the assessors will be asked to provide a guess as to which intervention the participant received and to disclose if the participant said which intervention they received.

Assessors

Trained and supervised assessors will carry out the consent, screening, and assessment procedures throughout Study Phase 1. The assessors will be recruited through Save the Children Sweden and receive a two-three day training on questionnaire administration, basic interviewing skills, common mental disorders, psychological first aid (PFA), and research ethics. There will be at least one assessor who is able to speak each language of the included participants. All assessors will be fluent in Swedish.

Sample Size

The primary aim of the feasibility RCT is to better understand the intervention and research procedures and is not intended to determine the effectiveness of the interventions. In turn, no power calculations have been carried out and the final sample size was based on previous feasibility trials of similar interventions, including the initial trials of Problem Management Plus A total number of 60 individuals, 20 per arm, will be included in the study which will allow us to evaluate the feasibility and acceptability of the PM+ and PM+EP interventions in Sweden.

Instruments

Assessment responses will be collected through REDcap, a digital medical research platform that will allow for the coding of questionnaires in multiple languages for ease of data collection and subsequent analysis.

Screening measures

The WHO Disability Assessment Schedule (WHODAS 2.0) socio-demographic and disability assessment questionnaires will both be collected at screening. The socio-demographic questionnaire will be used to collect information on age, gender, asylum status, marital status, education and work status, and living conditions. The WHODAS 2.0 is a questionnaire developed to measure health and disability corresponding to the following six domains: 1) cognition, 2) mobility, 3) self-care, 4) getting along, 5) life activities, and 6) participation. The 12-item version, which has been used more commonly as a screening-tool will be used to understand levels of impaired functioning. Scores are rated on a 1 (none) to 5 (extreme) scale (range: 12-60), with higher scores indicating worsened levels of functioning. A score of higher than 16 will be used to indicate decreased functionality. Minor adaptations of the questions have been made for this study to better suit youth; for example 'taking care of your household responsibilities?' was changed into 'Participating in household chores'. Community activities listed under item 4 (festivities, religious or other activities) were replaced with clubs, after school activities, religious or other activities.

The Kessler Psychological Distress Scale, 10-item version (K10) will be used to screen for levels of psychological distress. Items are scored on a scale of 1 (none of the time) to 5 (all of the time) with higher scores indicating higher levels of distress experienced in the preceding month (range 10 - 50). The K10 has been used extensively in adult populations and norms are available for young children aged 10 years old. Additionally, there are a number of studies that have validated the scale in adolescent populations. To align with other PM+ studies of refugees residing in HIC, we will use a cut-off score of 15 to indicate moderate levels of psychological distress.

Finally, imminent risk of suicide will be assessed using the three-item WHO PM+ suicide screener. The first question posed to participants is whether "in the past month have [they] had serious thoughts or a plan to end your life?". If the participant says no to this question the questionnaire will end and participants will be invited to participate in the trial dependent on their WHODAS 2.0 and K10 scores. If the participant says yes, two additional questions will be asked: (1) "Have you taken actions to end your life" and (2) "Do you plan to end your life in the next two weeks?". If the participant does not answer yes to these two questions they will be included in the study and this information will be flagged to their PM+ facilitator when providing support. If the participant does answer yes to any of the two additional questions, parents will be contacted for those under 18 years of age, and they will be referred to the emergency child psychiatric services immediately. If the parent is unable to assist the child and is not willing to accept further assistance, social services will be contacted. For adults older than 18 years of age, they will be referred to emergency psychiatric services. Transportation services will be contacted if needed.

Feasibility measures

The primary outcome of this study will be the feasibility and acceptability of the delivery of PM +EP in refugee youth. Feasibility will be decided on using the following criteria: a) 70% recruitment and consent rates, b) 70% attendance of sessions and assessments, c) 75% protocol adherence, d) maximum 10% presence of adverse events and no serious adverse events, e) fewer than 15% missing items on outcome measures, and f) qualitative assessments from the process evaluation.

Protocol adherence will be determined through two methods. The first is a self-rating fidelity checklist that will be filled out by the PM+/PM+EP facilitators at the end of each session. This will contain each of the elements from the completed session and facilitators will be asked to identify what items they completed and which items they may have missed to assess the degree of fidelity to the manualized intervention. Secondly, audio recordings of sessions will be taken if participants provide informed consent for recording. A random same of 10% of recordings will be scored independently by two research assistants. The interrater reliability for the audio recordings will be computed.

Secondary outcome measures

Secondary outcome measures will be administered at baseline and follow-up assessments to inform about possible effectiveness and preparation for a future definitive trial of PM+EP. The Hopkins Symptom Checklist-25 (HSCL-25) is a 25-item validated psychometric scale assessing symptoms of depression (15 items) and anxiety (10 items). Two of the depression items specifically relate to associated somatic symptoms. The items are rated on a 4-point Likert scale, ranging from 1 (not at all) to 4 (extremely) (range = 25-100). The measure has been often used in research including specifically with refugees and asylum seekers.

PTSD symptom severity, according to the DSM-5, will be established with the PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item checklist, corresponding to the 20 symptoms of PTSD as described in the DSM-5. Each item is scored on a 5-point scale scored from 0 (not at all) to 4 (extremely). When the symptom severity score is rated a two (moderate/threshold) or higher, a symptom is considered as present. Total symptom severity is calculated by summing the scores of the 20 items (range: 0-80), with higher scores indicating worsened severity of posttraumatic stress symptoms.

The Psychological Outcomes Profiles (PSYCHLOPS) will be used to indicate the client's perspective of change in their psychological distress level after therapy. The PSYCHLOPS has four questions measuring three domains; the problem(s) bothering the individual (two questions), how these problem(s) affect the daily functioning and wellbeing. Scores range from 0 to 5 and higher scores represent more psychological difficulty (range = 0-20).

Social support will be measured through a 1-item question assessing 'bonding social capital' from the Stockholm Public Health Cohort. Participants will be asked: "Do you know any people who can provide you with personal support for personal problems or crises in your life?". The response will be categorized as either high social support or low social support.

The Client Service Receipt Inventory (CSRI) will be used to track the health care services and medications that the participant has received in the three-months preceeding their entry to the study and over the course of the study.

To measure general well-being the World Health Organization 5-item Wellbeing Index (WHO-5) will be used. The questionnaire is a 5-item scale assessing general psychological wellbeing and quality of life as opposed to wellbeing tied to a certain psychopathology. Items are scored on a six-point scale ranging from 0 (at no time) to 5 (all of the time); total scores are the sum of the individual items with a range from 0 to 25. The scale has demonstrated sensitivity to change in well-being.

Lastly, the agency-subscale State Hope Scale (Adult version; SHS-A), will be used to measure hope among study participants. The agency-subscale of the SHS is a three-item scale measuring goal-directed behaviour during the intervention. Items are scored on an eight-point Likert scale ranging from 1 (definitely false) to 8 (definitely true). Total scores for agency are calculated by summing the item-level scores (range: 3-24). This measure will be translated into the relevant languages according to the WHO gold-standard guidelines on translation of psychological measures.

Other measures

Exposure to traumatic events will be assessed through a Traumatic Events Checklist (TEC). The checklist contains 23 forms of traumatic events that the participants may have experienced during their displacement and subsequent travel to Sweden. The checklist was developed and used among refugee populations residing in a number of contexts.

The Post-Migration Living Difficulties Checklist (PMLD) will be used to measure the level of post-migration challenges experienced by the participant during the last 12-months. The checklist contains 17-items measured on a five-point scale ranging from 0 (not a problem) to 4 (a very serious problem). Items that are either scored 3 or 4 are considered positive responses indicating a living difficulty. A total count of living difficulties is computer by summing the number of items scoring either a 3 or 4. For this study, three new items will be added to the list: (1) Bully or being rejected by peers, (2) Worries about future education and/or work, and (3) Arguments with parents over new friends and/or hobbies. Additional adaptations include adapting the item difficulties with employment to difficulties with education/employment, and adapting conflicts with social workers/other authorities to include teachers. The Ukrainian, Tigrinya and Arabic versions of the measure are available and Dari/Farsi translations will be made prior to the study.

Translation and adaptation of the measures

Where existing and validated translations of the above measures are not available, the WHO guidelines on the translations and adaptation of research instruments will be followed, which suggests the use of gold-standard guidelines on the translation of psychological measures. The methodology will be followed including forward- and back-translations by native speakers. Conflicting items will be discussed individually. Finally, cognitive interviews will be conducted to pilot-test the measures.

Interventions

Following the completion of the baseline assessment and randomization, all participants will receive an offer to attend a low-intensity psychological intervention, either PM+ (n=20) or PM+EP (n=20), or to receive CAU.

Problem Management Plus Problem Management Plus is a brief, potentially scalable psychological intervention developed by the World Health Organization and is delivered by non-specialised helpers. The intervention is described in detail elsewhere (Dawson et al., 2015). In brief, the intervention is based on cognitive behavioural therapy (CBT) techniques and typically consists of five weekly, ninety-minute sessions. Participants are taught the following techniques during the sessions: stress management, problem-solving, behavioural activation, and accessing social support. The effectiveness of both the individual and group formats of the PM+ intervention have been shown in a number of large definitive RCTs.

For the purposes of this study, an adapted version of PM+ will be used to match the exposure between the two active intervention arms. There will be six, weekly seventy-five-minute sessions as opposed to 5.

Problem Management Plus with Emotional Processing Module

To more directly address symptoms of traumatic stress, an adapted version of PM+ containing Emotional Processing module will be trialed in this study. The PM+ strategies discussed above are identical across both interventions apart from the additional module. The Emotional Processing module aims to provide a safe environment for participants to engage in the emotional processing of both positive and negative memories. During the additional session, participants will be asked to imagine significant memories as pieces of a jigsaw puzzle; participants will be asked to illicit three memories, two positive/pleasurable and one negative/frightening. Participants will be assisted in processing these memories through discussing the puzzle pieces, the thoughts and emotions that come with the memory, and future perspectives. Participants will be asked to rate the intensity of emotions before and after they talk about their memories each time they are brought up.

The additional module includes the following specific components:

1. Psychoeducation: Participants will be informed about the rationale behind the module and the mechanisms associated with it.
2. Choosing three pieces of their "jigsaw puzzle" (memories): Participants will be asked to choose three memories, two of them being pleasurable memories and one difficult (distressing/frightening/upsetting) memory. Participants will be asked to give a label to each of these memories (e.g. "leaving the country", "meeting with best friend").
3. Emotional processing of memories: After the "puzzle" is ready, participants will be asked to talk about the memories on their lifelines. Participants will be asked to first discuss the positive memory and then the difficult memory. Talking about the same difficult memory will last for three sessions. Each time it is discussed, a discussion about a positive memory will follow.
4. Positive imagination for the future: The final part of this module aims to help participants to engage in positive thinking by asking them to imagine their future in a positive way.

These components will occur between session three and session six. The PM+EP intervention will be six, weekly seventy-five-minute sessions.

Care as usual

The comparison group will receive care as usual (CAU) only. CAU for refugee youth (under 18) in Sweden corresponds to primary health care, education, social protection services, and specialized psychological treatment programs. However, adults are only able to access care that cannot be deferred. Once the individual has received their residence permit, they are able to access all healthcare. Upon first arriving in Sweden, refugees are referred to a municipality by the Swedish Board of Migration (Migrationsverket) until they have their residence permit. The municipality is responsible for education and social services while the regions are responsible for health care. In the regions, primary care is responsible for the first line of treatment but can also refer to the child and adolescent mental health services (CAMHS) if needed. Unaccompanied children might either be placed in families or in residential facilities and benefit from the same systems as accompanied children.

Save the Children, the implementing partner of this research has a large presence in providing care to children and youth with refugee backgrounds nationally. The care includes both psychosocial programming and three small mental health clinics for children. For this study, children will be recruited from the psychosocial programming. This involves for example youth groups, child-friendly spaces and after-school activities.

For this study, participants who are enrolled in specialized treatment programs at the screening phase will not be included in the study as they are receiving treatment, while PM+ aims to be preventative for the development of mental disorders for those who are psychologically distressed. However, when participants enroll in specialized mental health care during the study (i.e. after screening), they will not be excluded. In case participants use psychotropic medication at screening, they have to be on a stable dose for at least two months prior to enrollment in the study. If during the study's assessments participants receiving CAU show severe psychiatric disorders (e.g., psychosis) or risk of suicide that require specialist treatment and follow-up, they will be referred to an external specialist (e.g., psychiatrist).

Intervention helpers, trainers, and supervisors

Both the PM+ and PM+EP interventions will be delivered by helpers with at least a high school degree, matched to the participants according to their language and cultural backgrounds. The helpers will be native speakers of the language that the participant speaks and will also have sufficient speaking ability in Swedish or English. Where participants prefer, native Swedish speaking helpers will be available.

Prior to the study, helpers will receive a 9-day training that focuses on the PM+ strategies with additional training on common mental health problems, basic counseling skills, and self-care strategies. For those providing the PM+EP intervention, they will additionally be taught the Emotional Processing module. Following the training, helpers will be required to complete one practice case. Throughout their implementation of the intervention, helpers will receive supervision (either individual or group supervision).

PM+[EP] trainers and supervisors will be mental health professionals who have themselves received a five-day training of trainers (ToT). The ToT will be provided by a senior PM+ trainer and will include trainings on PM+ strategies and supervision skills. The PM+[EP] supervisors will receive regular supervision throughout the trial by a PM+ master trainer. Helpers, trainers, and supervisors will be primarily hired by Save the Children Sweden.

Participant Renumeration

Participants will not receive any direct renumeration for participation in the intervention itself to ensure that the treatment effects observed are attributable to the intervention and not financial gain. However, travel reimbursements will be made during the study for travel to and from the centres at which the interventions will be implemented (i.e. public transportation or standard fuel costs).

Participants will receive 200 SEK per assessment following intervention (1-week post-assessment, and 3-months follow-up assessment).

ELIGIBILITY:
Inclusion Criteria:

* 16 to 25 year old youth who arrived in Sweden in 2015 or later due to being forcibly displaced;
* Elevated levels of psychological distress as determined through the Kessler-10 psychological distress scale (K10; K10 > 15);
* Reduced levels of psychosocial functioning as measured by the WHO Disability Assessment Schedule (WHODAS 2.0; WHODAS 2.0 > 16);
* Assessment and manual are available in their preferred language, including Swedish.

Exclusion Criteria:

* An acute medical condition;
* Imminent suicide risk;
* Indication of psychotic disorders and substance-dependence;
* Indication of severe cognitive or neurological impairment;
* Receiving specialized mental health treatment;
* In case of current psychotropic medication used: change in dosage during the past two months.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability | From enrollment to the end of assessment prior (18 weeks)
  * 70% recruitment and consent rate
  * 70% attendance of sessions and assessments
  * 75% protocol adherence
  * Maximum 10% presence of adverse events and no serious adverse events
  * Fewer than 15% missing items on assessments

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS 2.0) | From enrollment to the end of assessment prior (18 weeks)
  Range: 0-48 Higher scores correspond to greater levels of disability
Hopkins Symptom Checklist-25 (HSCL-25) | From enrollment to the end of assessment prior (18 weeks)
  Range: 25-100 Higher total scores reflecting more severe anxiety and depression
PTSD Checklist for DSM-5 (PCL-5) | From enrollment to the end of assessment prior (18 weeks)
  Range: 0-80 Higher total scores indicate higher burden of posttraumatic stress symptoms
Self-identified problems (PSYCHLOPS) | From enrollment to the end of assessment prior (18 weeks)
Client Service Receipt Inventory | From enrollment to the end of assessment prior (18 weeks)
Bonding social capital | From enrollment to the end of assessment prior (18 weeks)
Subjective Wellbeing (WHO-5) | From enrollment to the end of assessment prior (18 weeks)
  Range: 0-25 Higher total scores reflecting higher levels of subjective wellbeing
State Hope Scale - Agency Subscale (SHS-A) | From enrollment to the end of assessment prior (18 weeks)
  Range: 0-21 Higher scores indicate higher levels of perceived agency
Post Migration Living Difficulties (PMLD) | From enrollment to the end of assessment prior (18 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum för stöd och behandling, Stockholm, Sweden

REFERENCES:
- [Derived] Mattelin E, Alozkan-Sever C, Shahnavaz S, Sijbrandij M, Mittendorfer-Rutz E, Akhtar A. Study Protocol of a feasibility and acceptability trial of Problem Management Plus with Emotional Processing (PM+EP) for forcibly displaced youth living in Sweden. BMJ Open. 2025 Oct 28;15(10):e104845. doi: 10.1136/bmjopen-2025-104845. PMID 41151965